CLINICAL TRIAL: NCT05293067
Title: Troponin in Carotid Revascularization
Acronym: TROPICAR
Status: Active, not recruiting | Type: Observational
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Igor Koncar, Vascular surgeon, MD, Ph.D., University of Belgrade
Other Study IDs: TROPICAR
Record Dates: First submitted 2022-03-04; First posted 2022-03-24 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A peripheral venous blood sample would be taken from all of the study participants in order to determine values of high-sensitive troponin. Troponin samples would be frozen and analyzed only after the patient's hospital discharge.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- carotid endarterectomy: High-sensitive troponin would be measured in patients undergoing carotid endarterectomy (CEA). Patients would be followed during the immediate postoperative period (until discharge from hospital), one month after, one and two years following the surgery, when researchers will gather information regarding the study outcomes during a regular postoperative control, or through telephone interviews.
  Interventions: Diagnostic Test: high-sensitive troponin
- carotid artery stenting: High-sensitive troponin would be measured in patients undergoing carotid artery stenting (CAS). Patients would be followed in the immediate postoperative period (until discharge from hospital), one month after, one and two years following the surgery, when researchers will gather information regarding the study outcomes during a regular postoperative control, or through telephone interviews.
  Interventions: Diagnostic Test: high-sensitive troponin

INTERVENTIONS:
Diagnostic Test: high-sensitive troponin — Values of high-sensitive troponin would be measured as follows: 1) preoperatively - one day before the planned intervention and 2) postoperatively - 8 hours after the operation and the first day after the operation.

SUMMARY:
Patients undergoing carotid revascularization procedures are at increased risk for the development of short- and long-term cardiac complications. Increased values of high-sensitive troponin may be useful in a timely selection of those patients. Still, contemporary literature doesn't provide enough data to answer the following questions: "Can high-sensitive troponin predict adverse cardiac outcomes perioperatively in carotid surgery?", "Should these cardiac biomarkers be routinely sampled in all patients undergoing carotid revascularization?" and "Can elevated levels of high-sensitive troponin preoperatively designate patients in whom the risk of surgical treatment (at a given moment) is greater than the benefit of the surgery?".

DETAILED DESCRIPTION:
The aims of the study are: 1) to determine the incidence of elevated troponin levels pre- and postoperatively in patients undergoing CEA/CAS; 2) to assess whether elevated troponin levels pre- and postoperatively can predict the occurrence of myocardial infarction and death in these patients; 3) to demonstrate whether routine pre- and postoperative troponin measurement is justified in all or only in a particular subpopulation of patients, and 4) to assess whether, in this regard, a difference between patients undergoing CEA and CAS procedures exists.

A prospective, multicenter cohort study would include approximately 240 consecutive patients undergoing CEA/CAS procedures, under the conditions of regional/general and local anesthesia, during the period from April, to August 2022. Patients admitted due to emergency procedure for immediate surgical treatment (the same day), patients with preoperative anemia (due to any reason, hemoglobin level < 10 g/dL), in whom concomitant or "staged" cardiac surgery or vascular procedure is planned, who had an acute coronary event in the previous 3 months, patients undergoing multiple CEA/CAS during the study period, as well as those patients with conditions that may lead to increased troponin levels (end-stage kidney disease, sepsis, acute pericarditis and myocarditis, advanced heart failure, chemotherapy, systemic inflammatory diseases, and critical limb ischemia) would be excluded from the study. Using a pre-designed questionnaire, standard demographic and clinical data (related to comorbidities, chronic therapy, habits, previous surgery, and characteristics of carotid disease) would be collected. Intraoperative data (type of carotid intervention, type of anesthesia technique, and shunt placement), as well as data regarding the postoperative course, would be obtained from the database implemented in daily practice and patients' medical records. High-sensitive troponin would be measured in all patients, according to the following plan: 1) preoperatively - one day before the planned intervention and 2) postoperatively - 8 hours after the operation and on the first day after the operation. Troponin samples would be frozen and analyzed only after the patient's hospital discharge. Also, ECG would be recorded immediately following troponin measurement (a day before the planned intervention, 8 hours and 24 hours after the intervention). Patients operated on at the Clinic for Vascular and Endovascular Surgery of the University Clinical Center of Serbia would be operated under the conditions of regional anesthesia - a combination of deep and superficial cervical plexus block (which is a regular practice at this Institution), or local infiltrative anesthesia (for CAS procedures), while patients in other Hospital would be treated under the conditions of general anesthesia (Collaborators - to be defined). Clinical outcomes of interest: myocardial injury, myocardial infarction, stroke, cardiac-related death, and the all-cause mortality, would be recorded perioperatively, until hospital discharge (2 days following the procedure). Myocardial infarction, stroke, cardiac-related death, and the all-cause mortality would be recorded preoperatively and up to 2 days following the procedure, one month after, one and two years following surgery (at regular postoperative check-ups or by telephone interview with the patient, or a member of his family). Myocardial injury would be defined in accordance with the current Fourth Universal Definition of Myocardial Infarction, published by the European Society of Cardiology, as the existence of at least one elevated troponin value above the 99th percentile of the upper reference limit. In accordance with the same recommendations, acute myocardial infarction would be defined as the existence of an increase and/or decrease in troponin levels and clinical signs of acute myocardial ischemia. The indication for surgery or stenting procedure would be made based on the European Society of Vascular Surgery guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Extracranial carotid stenosis greater than 50% (NASCET) in the carotid bifurcation or internal carotid artery assessed by ultrasound in whom carotid revascularisation is planned;
* The ability of the patient for follow-up examinations;
* Personally signed informed consent

Exclusion Criteria:

* Patients admitted due to emergency procedure for immediate surgical treatment (the same day);
* Patients with preoperative anemia (due to any reason, hemoglobin level < 10 g/dL);
* Patients in whom concomitant or "staged" cardiac surgery or vascular procedure is planned,
* Patients who had an acute coronary event in the previous 3 months;
* Patients undergoing multiple CEA/CAS during the study period;
* Patients with end-stage kidney disease;
* Patients with sepsis:
* Patients with acute pericarditis/myocarditis;
* Patients with advanced heart failure;
* Patients on chemotherapy,
* Patients with systemic inflammatory diseases;
* Patients with critical limb ischemia;

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with extracranial carotid stenosis greater than 50% (NASCET) in the carotid bifurcation or internal carotid artery assessed by ultrasound in whom carotid revascularisation is planned;
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of myocardial injury | preoperatively
  Myocardial injury would be defined in accordance with the current Fourth Universal Definition of Myocardial Infarction, published by the European Society of Cardiology, as the existence of at least one elevated troponin value above the 99th percentile of the upper reference limit.
The incidence of myocardial injury | 2 days following surgery
  Myocardial injury would be defined in accordance with the current Fourth Universal Definition of Myocardial Infarction, published by the European Society of Cardiology, as the existence of at least one elevated troponin value above the 99th percentile of the upper reference limit.
The incidence of myocardial infarction | 2nd postoperative day
  Myocardial infarction would be defined as the existence of an increase and/or decrease in troponin levels and clinical signs of acute myocardial ischemia, in accordance with the Fourth Universal Definition of Myocardial Infarction.
The incidence of myocardial infarction | 2 years following surgery
  Myocardial infarction would be defined as the existence of an increase and/or decrease in troponin levels and clinical signs of acute myocardial ischemia, in accordance with the Fourth Universal Definition of Myocardial Infarction.
The rate of cardiac-related death | 2nd postoperative day
  Cardiac-related death would be defined as any lethal outcome that resulted due to progression of heart disease.
The rate of cardiac-related death | 2 years following surgery
  Cardiac-related death would be defined as any lethal outcome that resulted due to progression of heart disease.
The incidence of stroke | 2nd postoperative day
  Stroke would be defined as rapidly developing clinical signs of focal (or global) disturbance of cerebral function, lasting more than 24 hours or leading to death, with no apparent cause other than that of vascular origin, with the evidence of acute infarction on brain computed tomography or magnetic resonance imaging.
The incidence of stroke | 2 years following surgery
  Stroke would be defined as rapidly developing clinical signs of focal (or global) disturbance of cerebral function, lasting more than 24 hours or leading to death, with no apparent cause other than that of vascular origin, with the evidence of acute infarction on brain computed tomography or magnetic resonance imaging.
The rate of all-cause mortality | 2nd postoperative day
  All-cause mortality would refer to any lethal outcome (due to any cause), that would occur during the study.
The rate of all-cause mortality | 2 years following surgery
  All-cause mortality would refer to any lethal outcome (due to any cause), that would occur during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Koncar, MD, Ph.D., Principal Investigator — University of Belgrade
Locations (1):
- Clinic for Vascular and Endovascular Surgery, University Clinical Center of Serbia, Belgrade, Serbia, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grobben RB, Vrijenhoek JE, Nathoe HM, Den Ruijter HM, van Waes JA, Peelen LM, van Klei WA, de Borst GJ. Clinical Relevance of Cardiac Troponin Assessment in Patients Undergoing Carotid Endarterectomy. Eur J Vasc Endovasc Surg. 2016 Apr;51(4):473-80. doi: 10.1016/j.ejvs.2015.09.023. Epub 2015 Nov 6. PMID 26553374
- [Background] Galyfos G, Tsioufis C, Theodorou D, Katsaragakis S, Zografos G, Filis K. Cardiac troponin I after carotid endarterectomy in different cardiac risk patients. J Stroke Cerebrovasc Dis. 2015 Mar;24(3):711-7. doi: 10.1016/j.jstrokecerebrovasdis.2014.11.024. Epub 2015 Jan 16. PMID 25601178
- [Background] Pereira-Macedo J, Rocha-Neves JP, Dias-Neto MF, Andrade JPV. Prognostic effect of troponin elevation in patients undergoing carotid endarterectomy with regional anesthesia - A prospective study. Int J Surg. 2019 Nov;71:66-71. doi: 10.1016/j.ijsu.2019.09.015. Epub 2019 Sep 19. PMID 31542388
- [Background] Nagy B, Engblom E, Matas M, Maroti P, Koszegi T, Menyhei G, Lantos J, Szabo P, Molnar T. Increased serum level of high sensitivity troponin T even prior to surgery can predict adverse events during carotid endarterectomy. Vascular. 2021 Dec;29(6):938-944. doi: 10.1177/1708538120986297. Epub 2021 Jan 11. PMID 33427096